CLINICAL TRIAL: NCT02989467
Title: A Single-Center, Placebo-Controlled, Double-Blind Study to Evaluate the Effects of Aprepitant on Satiation, Gastric Volume, Gastric Accommodation and Gastric Emptying in Healthy Volunteers
Brief Title: Effects of Aprepitant on Satiation, Gastric Volume, Gastric Accommodation and Gastric Emptying
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Professor, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-007929
Record Dates: First submitted 2016-12-07; First posted 2016-12-12 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Healthy
MeSH Terms: interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aprepitant (Active Comparator): Subjects will receive one tablet daily for 5 consecutive days. On Day 1 subjects will take a 125mg tablet, on Days 2-5, subjects will take an 80 mg tablet.
  Interventions: Drug: Aprepitant
- Placebo (Placebo Comparator): Subjects will receive one placebo tablet daily for 5 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant — Subjects will receive one tablet daily for 5 consecutive days. On Day 1 subjects will take a 125mg tablet, on Days 2-5, subjects will take an 80 mg tablet.
  Other Names: Emend
  Arms: Aprepitant
Drug: Placebo — Subjects will receive one placebo tablet daily for 5 consecutive days.
  Arms: Placebo

SUMMARY:
This research study is being done to compare the effects of Aprepitant and placebo on fasting gastric volume, accommodation volume, satiation (fullness) and gastric emptying.

ELIGIBILITY:
Inclusion criteria:

1. Able to provide written consent
2. No medical problems or chronic diseases, specifically, no type 2 diabetes mellitus
3. Body Mass Index of 18-35 kg/m^2
4. Female subjects must have negative urine pregnancy tests and must not be lactating prior to receiving study medication and radiation exposure
5. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study
6. Female subjects unable to bear children must have this documented in the medical record (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period])

Exclusion criteria:

1. Diagnosis of gastrointestinal diseases
2. Structural or metabolic diseases that affect the gastrointestinal system
3. Unable to avoid the following over-the-counter medications 48 hours prior to the baseline period and throughout the study:

   * Medications that alter GI transit including laxatives, magnesium and aluminum containing antacids, prokinetics, erythromycin
   * Analgesic drugs including NSAIDs and cyclooxygenase-2 (COX-2) inhibitor. (NOTE: Stable doses of thyroid replacement, estrogen replacement, low-dose aspirin for cardioprotection, and birth control (but with adequate backup contraception as drug-interactions with birth control have not been conducted) are permissible.)
4. History of recent surgery (within 60 days of screening).
5. Acute or chronic illness or history of illness, which in the opinion of the investigator could pose a threat or harm to the subject or obscure interpretation of laboratory test results or interpretation of study data such as frequent angina, Class III or IV congestive heart failure, moderate impairment of renal or hepatic function, poorly controlled diabetes, etc.
6. Any clinically significant abnormalities on physical examination or laboratory abnormalities identified in the medical record, as determined by the investigator.
7. Acute GI illness within 48 hours of initiation of the baseline period.
8. Females who are pregnant or breastfeeding.
9. History of excessive alcohol use or substance abuse.
10. Participation in an investigational study within the 30 days prior to dosing in the present study.
11. Any other reason, which in the opinion of the investigator would confound proper interpretation of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Gastric Emptying Half-Time of Solids as Measured by Scintigraphy | Day 3, approximately 2 hours after radiolabeled meal is ingested
  The time for half of the ingested solids to leave the stomach.
Satiation Expressed as Volume to Fullness | Day 4, approximately 30 minutes after liquid meal
  Subjects will do a satiation/nutrient drink test, consuming Ensure at a relatively constant rate of 30 ml/min. Subjects will record their sensations every 5 minutes using a numerical scale from 0-5, with level 0 being no symptoms, level 3 corresponding to fullness sensation after a typical meal, and level 5 corresponding to the maximal tolerated volume (maximum or unbearable fullness/satiation). This measure is the volume consumed when the fullness sensation reaches level 3.
Fasting Gastric Volume as Measured by Single Photon Emission Computed Tomography (SPECT) | Day 5, approximately 15 minutes after radioactive marker is administered
  Subjects will arrive to the Clinical Research and Trials Unit (CRTU) fasting. A radioactive marker will be administered intravenously. After a 10-15 minute wait period a fasting scan will be acquired using a dual-head gamma camera.
Postprandial Gastric Volume as Measured by SPECT | Day 5, approximately 30 minutes after liquid meal
  At the completion of the fasting scan, the subject will consume 300 ml of Ensure followed by a postprandial scan using a dual-head gamma camera.
Accommodation Volume as Measured by SPECT | Day 5, approximately 30 minutes after liquid meal
  This variable is calculated as postprandial gastric volume minus fasting volume.

SECONDARY OUTCOMES:
Solid Gastric Emptying: Proportion of Meal Emptied at 2 Hours | Day 3, approximately 2 hours after radiolabeled meal is ingested
  On Day 3, subjects will take part in a gastric emptying by scintigraphy test. Subjects will be given a scrambled egg breakfast with toast and a glass of milk. The eggs and milk contain a small amount of radioactive substance. At the completion of the meal, subjects will stand in front of a special camera and pictures were taken at specific intervals. This outcome measure is the proportion of the radiolabeled meal emptied at 2 hours.
Solid Gastric Emptying: Proportion of Meal Emptied at 4 Hours | Day 3, approximately 4 hours after radiolabeled meal is ingested
  On Day 3, subjects will take part in a gastric emptying by scintigraphy test. Subjects will be given a scrambled egg breakfast with toast and a glass of milk. The eggs and milk contain a small amount of radioactive substance. At the completion of the meal, subjects will stand in front of a special camera and pictures were taken at specific intervals. This outcome measure is the proportion of the radiolabeled meal emptied at 4 hours.
Maximum Tolerated Volume on Satiation Test | Day 4, approximately 30 minutes after liquid meal
  On Day 4, subjects will do a satiation/nutrient drink test. Participants will record their sensations every 5 minutes using a numerical scale from 0-5, with level 0 being no symptoms, level 3 corresponding to fullness sensation after a typical meal, and level 5 corresponding to the maximal tolerated volume (maximum or unbearable fullness/satiation). This measure is the volume consumed when the fullness sensation reaches level 5.
Individual Symptom Scores (Nausea, Bloating, Fullness, Pain) on Satiation Test | Day 4, approximately 30 minutes after liquid meal
  Postprandial symptoms of nausea, bloating, fullness, and pain will be measured using 100 mm horizontal visual analog scales, with the words "none" and "worst ever" anchored at each end.
Aggregate Symptoms Score | Day 4, approximately 1 hour after liquid meal
  Postprandial symptoms of nausea, bloating, fullness, and pain will be measured using 100 mm horizontal visual analog scales, with the words "none" and "worst ever" anchored at each end. The aggregate symptoms score is calculated by adding the mean individual scores. The lowest possible score would be 0 (none) and the highest maximum score possible is 400 (worst ever).
Gastric Volume Ratio | Day 5, approximately 1 hour after radioactive marker is administered
  Postprandial/fasting gastric volume
Absolute postprandial gastric volume | Day 5, approximately 1 hour after radioactive marker is administered
  This is the total postprandial gastric volume

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided